# A prospective, double-blind, randomized pilot study evaluating the effects of Toradol versesplacebo for pain control after donor nephrectomy.[820]

Principal Investigator: Jeffrey Campsen/Eddie Martinez

SAP Author: Angela P. Presson Project Lead: Chelsea Allen Additional Statistician(s):

Date: 10/31/2017

#### Introduction

This is a randomized controlled trial (RCT) comparing placebo to toradol treatment for pain control after donor nephrectomy. The primary outcomes of interest include narcotic use and length of stay (LOS), where the hypothesis is that toradol will reduce post-operative narcotic use and LOS. The study was powered on the safety outcome allowing for a limited creatinine increase on post-operative day 1. The rationale being that regardless of toradol efficacy, if it was not safe to use then it would not be adopted into clinical practice.

### Investigator's Description

Completed pilot study now need power calculation for a prospective, double-blind, randomized pilot study evaluating the effects of Toradol, and Lyrica verses placebo for pain control after donor nephrectomy.

# **Project Endpoints**

Paper, ASTS abstract 11/22/17

#### Data

The raw data set is at: Campsen\_Jeffrey\_820\_toradol\_rct\Data\Raw\Torpedo II Study.xlsx, the analysis data set is: Campsen\_Jeffrey\_820\_toradol\_rct\Data\Torpedo II Study - Recoded.xlsx.

#### **Exposure Variables**

The variable "group" in the analysis data set describes the exposure group, toradol versus placebo.

#### <u>Outcomes</u>

cr.ratio = Construct this safety outcome of fold change in creatinine within the toradol group (pre-op/post op day 1), constructed from the variables cr.pre and cr.pod1.

cum.me = The post-operative narcotic usage outcome in morphine equivalents (ME).

postop.los = Hospital LOS.

#### Inclusion/Exclusion

None, all patients in the data set were included in the analysis

## **Research Objectives**

- 1. Compare patient characteristics: age, height, weight, bmi, sex, race, operative time, side, opioid usage, hct pre, hct pacu, hct pod1, hct diff, hct ratio, cr pre, cr pod1, cr ratio, postop nausea, failed foley and postop LOS between toradol and control groups.
- 2. Assess the creatinine safety outcome using a non-inferiority test that the fold change is at most two-fold, or alternatively for the pre-surgery creatinine group to be ≥0.5 times the post-surgery.

## **Analyses**

For the comparison of patient characteristics, we will use the R functions developed by our center to implement simple statistical tests selected from the following options: 1=t.test, 2=Wilcox, 3=Chi-square, 4=Fisher's exact, 5=Fisher's exact test with simulation, 6=Exact wilcoxon rank sum test. The following table indicates our results and which test was used for which variable.

Table 1. Summary by group.

| placebo (N=29) | Toradol (N=33) | P-value | Test |
|---|---|---|---|
| 45.1 (12.2) | 43.8 (11) | 0.68 | 1 |
| 44 (35, 53) | 42 (34, 52) | - | - |
| (26, 69) | (25, 66) | - | - |
| | 169.9 (9.4) | 0.47 | 1 |
| 170.2 (166.4, 179) | 170.2 (162.6, 172.7) | - | - |
| (154.9, 190.5) | (156, 195.6) | - | - |
| 79.6 (13.3) | 77.7 (16.3) | 0.62 | 1 |
| 80.3 (70.5, 88.9) | 77.4 (64.5, 88) | - | - |
| (56.2, 109) | (50.9, 123) | - | - |
| 26.9 (3.2) | 26.6 (4.7) | 0.76 | 1 |
| 27.3 (24, 28.9) | 27.5 (22.1, 30) | - | - |
| (21, 33.4) | (17.1, 34.8) | - | - |
| 17 (59%) | 26 (79%) | 0.086 | 3 |
| 12 (41%) | 7 (21%) | - | - |
| 0 (0%) | 1 (3%) | 0.4 | 4 |
| 0 (0%) | 1 (3%) | - | - |
| 3 (10%) | 1 (3%) | - | - |
| 26 (90%) | 29 (91%) | - | - |
| 2 (7%) | 2 (6%) | >0.99 | 4 |
| 27 (93%) | 29 (94%) | - | - |
| 129.3 (30) | 124.7 (27.8) | - | - |
| 124 (110, 135) | 116 (110, 128) | 0.33 | 6 |
| (80, 200) | (99, 245) | - | - |
| 20 (69%) | 25 (76%) | 0.55 | 3 |
| 9 (31%) | 8 (24%) | - | - |
| 62.9 (65.2) | 31.1 (25.5) | - | - |
| 45 (25, 70.8) | 27 (13, 42.3) | 0.006 | 6 |
| | 45.1 (12.2)<br>44 (35, 53)<br>(26, 69)<br>171.6 (8.9)<br>170.2 (166.4, 179)<br>(154.9, 190.5)<br>79.6 (13.3)<br>80.3 (70.5, 88.9)<br>(56.2, 109)<br>26.9 (3.2)<br>27.3 (24, 28.9)<br>(21, 33.4)<br>17 (59%)<br>12 (41%)<br>0 (0%)<br>0 (0%)<br>3 (10%)<br>26 (90%)<br>2 (7%)<br>27 (93%)<br>129.3 (30)<br>124 (110, 135)<br>(80, 200)<br>20 (69%)<br>9 (31%)<br>62.9 (65.2) | 45.1 (12.2) | 45.1 (12.2) 43.8 (11) 0.68 44 (35, 53) 42 (34, 52) - (26, 69) (25, 66) - 171.6 (8.9) 169.9 (9.4) 0.47 170.2 (166.4, 179) 170.2 (162.6, 172.7) - (154.9, 190.5) (156, 195.6) - 79.6 (13.3) 77.7 (16.3) 0.62 80.3 (70.5, 88.9) 77.4 (64.5, 88) - (56.2, 109) (50.9, 123) - 26.9 (3.2) 26.6 (4.7) 0.76 27.3 (24, 28.9) 27.5 (22.1, 30) - (21, 33.4) (17.1, 34.8) - 17 (59%) 26 (79%) 0.086 12 (41%) 7 (21%) - 0 (0%) 1 (3%) - 3 (10%) 1 (3%) - 2 (90%) 29 (91%) - 2 (7%) 2 (6%) >0.99 27 (93%) 29 (94%) - 124 (110, 135) 116 (110, 128) 0.33 (80, 200) (99, 245) - 20 (69%) 25 (76%) 0.55 9 (31%) 8 (24%) |

| Variable* | placebo (N=29) | Toradol (N=33) | P-value | Test |
|---|---|---|---|---|
| -Range | (10.7, 343.8) | (0.7, 111) | - | - |
| hct.pre - Mean (SD) | 44.1 (2.8) | 43.5 (3) | 0.4 | 1 |
| -Median (IQR) | 44.5 (42.1, 45.6) | 43.1 (41.5, 44.8) | - | - |
| -Range | (38.3, 51) | (38.7, 50) | - | - |
| hct.pacu - Mean (SD) | 41.8 (3.4) | 39.9 (3.2) | 0.023 | 1 |
| -Median (IQR) | 42.2 (39.4, 44.3) | 39.5 (38.3, 40.8) | - | - |
| -Range | (34.9, 47) | (34.4, 48.3) | - | - |
| hct.pod1 - Mean (SD) | 39.8 (3.5) | 37.2 (2.7) | 0.002 | 1 |
| -Median (IQR) | 40.1 (37.5, 42.4) | 36.9 (35.9, 38.2) | - | - |
| -Range | (33.6, 45.7) | (32.6, 46.3) | - | - |
| hct.diff - Mean (SD) | 4.3 (2.5) | 6.3 (2.1) | 0.002 | 1 |
| -Median (IQR) | 4.7 (2.5, 5.7) | 6.4 (5, 7.3) | - | - |
| -Range | (-1.9, 9.5) | (1.7, 12.5) | - | - |
| hct.ratio - Mean (SD) | 1.1 (0.1) | 1.2 (0.1) | < 0.001 | 1 |
| -Median (IQR) | 1.1 (1.1, 1.2) | 1.2 (1.1, 1.2) | - | - |
| -Range | (1, 1.3) | (1, 1.3) | - | - |
| cr.pre - Mean (SD) | 0.9(0.1) | 0.8(0.2) | 0.65 | 1 |
| -Median (IQR) | 0.9(0.8, 0.9) | 0.8(0.7, 0.9) | <u>-</u> | <u>-</u> |
| -Range | (0.6, 1.1) | (0.6, 1.2) | <mark>-</mark> | _ |
| cr.pod1 - Mean (SD) | 1.3 (0.3) | 1.3 (0.3) | 0.87 | _ 1 |
| -Median (IQR) | 1.2 (1.1, 1.5) | 1.2 (1.1, 1.4) | <u>-</u> | _ |
| -Range | (0.8, 1.9) | (0.9, 1.9) | <mark>-</mark> | _ |
| cr.ratio - Mean (SD) | 0.7(0.1) | 0.6(0.1) | 0.19 | _ 1 |
| -Median (IQR) | 0.7(0.6, 0.7) | 0.6(0.6, 0.7) | <u>-</u> | |
| -Range | (0.5, 1) | (0.5, 0.8) | _ | _ |
| postop.nasea -N | 5 (17%) | 8 (24%) | 0.5 | 3 |
| Y | 24 (83%) | 25 (76%) | - | - |
| failedfoley -N | 29 (100%) | 32 (97%) | >0.99 | 4 |
| Y | 0 (0%) | 1 (3%) | - | - |
| postop.los -Mean (SD) | 56.1 (16) | 50 (13.5) | - | _ |
| -Median (IQR) | 57.3 (50.6, 66.3) | 51.5 (46.5, 56) | 0.029 | 6 |
| -Range | (26.4, 82.2) | (23.6, 81.1) | - | _ |

<sup>\*</sup>Missing values: race =1, ethnicity =2,

Test: 1=t.test, 2=Wilcox, 3=Chi-square, 4=Fisher's exact, 5=Fisher's exact test with simulation, 6=Exact wilcoxon rank sum test

2. The safety analysis was conducted using a 1-sided t-test compared to a 0.5 fold change. Here are the results:

A one-sided t-test shows that the pre-surgery creatinine increase over the post-surgery measure  $\left(\frac{\text{HCT Pre-OP}}{\text{HCT Post-OP Day 1}}\right)$  within the Toradol group has a mean fold change of 0.64 (95% CI: 0.62, 0.66), which is over the safety level of a 0.5 fold change (because this is pre/post). The p-value for this test is less than 0.0001, thus the Toradol group meets the safety threshold.

#### **Power Calculation**

The primary safety outcome is defined by a creatinine increase on post-operative day 1 of at most 100% (ie, twice the pre surgery measure) in the toradol group. To achieve 90% power at a 2.5% significance level for testing that the post-surgery creatinine increase is at most two-fold (where 1.5 fold is expected), or alternatively for the pre-surgery creatinine group to be  $\geq$ 0.5 times the post-surgery, we need 17 subjects in the toradol group. This calculation was based on a non-inferiority test (one sided t-test).

# **Quality Control (QC) Plans**

The analysis plan and code was reviewed by two independent statisticians.

# **SDBC Information**

Please remember to acknowledge the SDBC: "This investigation was supported by the University of Utah Study Design and Biostatistics Center, with funding in part from the National Center for Research Resources and the National Center for Advancing Translational Sciences, National Institutes of Health, through Grant 8UL1TR000105 (formerly UL1RR025764)."



The University of Utah
Study Design and Biostatistics Center
Center for Clinical and Translational Science
<a href="http://www.ccts.utah.edu/biostats/">http://www.ccts.utah.edu/biostats/</a>